CLINICAL TRIAL: NCT00295347
Title: Mineralocorticoid Receptor in the Treatment of Severe Depression: A Randomized, Double Blind, and Placebo Controlled Trial
Brief Title: Mineralocorticoid Receptor in the Treatment of Severe Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OT 209/3-1
Record Dates: First submitted 2006-02-22; First posted 2006-02-23 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Spironolactone; Fludrocortisone; Escitalopram

INTERVENTIONS:
Drug: Spironolactone
Drug: fludrocortisone
Drug: escitalopram

SUMMARY:
The proposed research aims to compare the onset of action and the efficacy of fludrocortisone, a mineralocorticoid receptor agonist vs. spironolactone, a mineralocorticoid antagonist, vs. placebo as augmentation to a selective serotonin reuptake inhibitor (SSRI) in 65 inpatients with severe depression. The study will also explore the utility of the hypothalamic-pituitary-adrenal (HPA) axis in predicting treatment response. The study will be a 5-week randomized and double-blind trial of fludrocortisone vs. spironolactone vs. placebo during three years.

ELIGIBILITY:
Inclusion Criteria:

* Depressed male and female inpatients according to DSM-IV
* Age between 18 and 70 years
* Minimum of 17-items Hamilton Depression Score of 18
* Informed consent signed

Exclusion Criteria:

* Relevant medical or neurological disorders
* Pregnancy or unsure contraception
* Relevant psychiatric comorbidity
* Active alcohol or other substance abuse/dependance
* Contraindications to SSRI, fludrocortisone, or spironolactone
* Steroid medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Otte, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany